CLINICAL TRIAL: NCT03863977
Title: Comparison of Post-operative Analgesic Effects of Two Doses of Dexamethasone Added to Bupivacaine in Ultrasound-guided Transversusabdominis Plane (TAP) Block for Inguinal Hernia Repair
Brief Title: Post-operative Analgesic Effects of Dexamethasone Added to Bupivacaine in Transversusabdominis Plane (TAP) Block
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amani Hassan Abdel-Wahab, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB:17100670
Record Dates: First submitted 2019-03-03; First posted 2019-03-05 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Postoperative Analgesia
Keywords: TAP block; inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Dexamethasone; dexamethasone acetate; Bupivacaine

STUDY DESIGN:
Intervention Model Description: 60 patients will be divided into two groups according to the dose of dexamethasone added to bupivacaine in the TAP block, I - group ( Group D4 ) 4mg of dexamethasone will be added II - group ( Group D8 ) 8mg of dexamethasone will be added. III-group(control) bupivacaine alone
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A blinded physician prepared the study medications in color coded syringes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dex4 group (Active Comparator): After the surgery, the patients in this group will receive 4 mg dexamethasone added to 1mg/kg of 0.5% bupivacaine in the TAP block.
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine
- Dex8 group (Active Comparator): After the surgery, the patients in this group will receive 8 mg dexamethasone added to 1mg/kg of 0.5% bupivacaine in the TAP block.
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine
- control group (Active Comparator): After the surgery, the patients in this group will 1mg/kg of 0.5% bupivacaine in the TAP block.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexamethasone — After the surgery, dexamethasone added to 1mg/kg of 0.5% bupivacaine in the TAP block.
  Other Names: dexamethasone acetate
  Arms: Dex4 group; Dex8 group
Drug: Bupivacaine — After the surgery,1mg/kg of 0.5% bupivacaine in the TAP block.
  Other Names: plain marcaine

SUMMARY:
To compare the postoperative analgesic effect of two doses of dexamethasone added to bupivacaine in ultrasound-guided TAP block for inguinal hernia repair.

DETAILED DESCRIPTION:
The transverses abdominis plane block (TAP block) is a regional anesthesia technique that provides analgesia following abdominal surgery . The TAP block significantly reduces pain after open inguinal hernia repair, regardless of whether it is used as a primary anesthesia technique or as a complement to general anesthesia, spinal or local anesthesia .

The investigators designed this study to compare the postoperative analgesic effect of two doses of dexamethasone( 4 mg and 8 mg ) added to bupivacaine in ultrasound-guided TAP block for inguinal hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age from 18 to 60 years old,
* physical status ASA I-II (by the American Society of Anesthesiologists),
* Elective unilateral open inguinal hernia repair,
* Under spinal anesthesia

Exclusion Criteria:

* age < 18 or > 60,
* American society of anesthesiologist (ASA)class III-IV,
* known allergy to amino amide local anesthetics,
* skin infection and diseases at site of injection.
* coagulation disorders,
* patients with body mass index (BMI) > 35 kg/m2,
* scrotal hernias,

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
time of the first analgesic request | in the first postoperative 24 hours
  time of the first analgesic request in the first postoperative 24 hours ,patients will receive analgesia if visual analog scale (VAS) score more than 3

SECONDARY OUTCOMES:
change in visual analog scale (VAS) | 2nd, 4th, 8th, 16th, and 24th postoperative hours.
  measuring the change in visual analog scale VAS (0: no pain to 10: worst imaginable pain), to evaluate postoperative analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Amany Hassan, Lectural, Principal Investigator — Assiut university, Egypt
Locations (1):
- Assiut university hospitals, Asyut, Assiut Governorate, Egypt